CLINICAL TRIAL: NCT01305291
Title: Fibersol-2 Clinical Trials Related to Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: Archer Daniels Midland Co. (Industry)
Responsible Party: Suzanne Hendrich, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ADM FB2-1 Hendrich; 08-291 (Other: ISU IRB)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Lack of Satiety
Keywords: dietary fiber; satiety response; hunger; CCK; PYY; ghrelin; GIP; GLP-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- tea only without fibersol-2 (Placebo Comparator): * On the day before the test, subjects need to consume their evening meal before 9 pm, and fast until the start of the test the next day.
  * The evening meal will be a standardized meal for all subjects (11).
  * They are allowed to consume water up until 1 hr before the test.
  * Before the start of the test a cannula will be inserted into the ante-cubital arm vein for use of repeated blood sampling (11).
  * The beverage will be consumed at 10 am.
  * Blood samples will be taken at specified time points prior to after the treatments.
  Interventions: Other: placebo
- tea only with fibersol-2 (10 g) (Active Comparator): * On the day before the test, subjects need to consume their evening meal before 9 pm, and fast until the start of the test the next day.
  * The evening meal will be a standardized meal for all subjects.
  * They are allowed to consume water up until 1 hr before the test.
  * Before the start of the test a cannula will be inserted into the ante-cubital arm vein for use of repeated blood sampling (11).
  * The beverage will be consumed at 10 am.
  * Blood samples will be taken at specified time points prior to and after the treatments.
  * Ingredient only test will be done without the meal to determine independent effects of Fibersol-2.
  Interventions: Dietary Supplement: digestion-resistant maltodextrin
- tea without fibersol-2 and meal (Placebo Comparator): * On the day before the test, subjects need to consume their evening meal before 9 pm, and fast until the start of the test the next day.
  * The evening meal will be a standardized meal for all subjects.
  * They are allowed to consume water up until 1 hr before the test.
  * Before the start of the test a cannula will be inserted into the ante-cubital arm vein for use of repeated blood sampling.
  * The test meal and beverage will be consumed at 10 am.
  * The meal will consist of pasta meal (main pasta dish = Carb 64.5%, Fat 17.7%, Protein 17.8%; total kcal 739).
  * Tea containing test materials will accompany the meal.
  * Blood samples will be taken at specified time points prior to and after the treatments.
  Interventions: Other: placebo
- tea with 5 g fibersol-2 and meal (Experimental): * On the day before the test, subjects need to consume their evening meal before 9 pm, and fast until the start of the test the next day.
  * The evening meal will be a standardized meal for all subjects.
  * They are allowed to consume water up until 1 hr before the test.
  * Before the start of the test a cannula will be inserted into the ante-cubital arm vein for use of repeated blood sampling.
  * The test meal and beverage will be consumed at 10 am.
  * The meal will consist of pasta meal (main pasta dish = Carb 64.5%, Fat 17.7%, Protein 17.8%; total kcal 739).
  * Tea containing test materials will accompany the meal.
  * Blood samples will be taken at specified time points prior to and after the treatments.
  Interventions: Dietary Supplement: digestion-resistant maltodextrin
- tea with 10 g fibersol-2 and meal (Experimental): * On the day before the test, subjects need to consume their evening meal before 9 pm, and fast until the start of the test the next day.
  * The evening meal will be a standardized meal for all subjects.
  * They are allowed to consume water up until 1 hr before the test.
  * Before the start of the test a cannula will be inserted into the ante-cubital arm vein for use of repeated blood sampling.
  * The test meal and beverage will be consumed at 10 am.
  * The meal will consist of pasta meal (main pasta dish = Carb 64.5%, Fat 17.7%, Protein 17.8%; total kcal 739).
  * Tea containing test materials will accompany the meal.
  * Blood samples will be taken at specified time points prior to and after the treatments.
  Interventions: Dietary Supplement: digestion-resistant maltodextrin

INTERVENTIONS:
Other: placebo
  Arms: tea only without fibersol-2; tea without fibersol-2 and meal
Dietary Supplement: digestion-resistant maltodextrin
  Other Names: Fibersol-2
  Arms: tea only with fibersol-2 (10 g); tea with 10 g fibersol-2 and meal; tea with 5 g fibersol-2 and meal

SUMMARY:
Emerging research suggests fiber, particularly digestion-resistant maltodextrins such as Fibersol-2, may impact satiety, by decreasing hunger, prolonging satiation, and/or increasing satiety signals from the gut. This research aims to determine whether or not Fibersol-2 may impact satiety, by decreasing hunger, prolonging satiation, and/or increasing satiety signals from the gut.

ELIGIBILITY:
Inclusion Criteria:

i. No known food allergies

ii. Normal healthy individuals

iii. No food intake abnormalities or abnormal feeding behaviors

iv. Average American BMI (21-28)

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Visual analog scale questionnaire subjective satiety responses | 4 hours
  Hunger survey (30 minutes before meal and every half hour for 4 hours postprandial) (analogue scores)
serum cholecystokinin (CCK) | 4 hours
  0, 30, 60, 120, 180, and 240 min post-meal
serum peptide YY (PYY) | 4 hours
  0, 30, 60, 120, 180, and 240 min post-meal
serum glucagon-like peptide-1 (GLP-1) | 4 hours
  0, 30, 60, 120, 180, and 240 min post-meal
serum ghrelin | 4 hours
  0, 30, 60, 120, 180, and 240 min post-meal
serum gastric inhibitory peptide (GIP) | 4 hours
  0, 30, 60, 120, 180, and 240 min post-meal

SECONDARY OUTCOMES:
serum total cholesterol | 4 hours
  0, 30, 60, 120, 180, 240 min
serum LDL-cholesterol | 4 hours
  0, 30, 60, 120, 180, 240 min
serum HDL-cholesterol | 4 hours
  0, 30, 60, 120, 180, 240 min
serum triglycerides | 4 hours
  0, 30, 60, 120, 180, 240 min
serum free fatty acids | 4 hours
  0, 30, 60, 120, 180, 240 min
serum glucose | 2 hours
  0, 30, 60, 90, 120 min
serum insulin | 2 hours
  0, 30, 60, 90, 120 min
gastrointestinal symptoms questionnaire | 24 h
  subjects recorded incidents and severity of gastrointestinal symptoms post treatment over 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hendrich, PhD, Principal Investigator — Iowa State University
Locations (1):
- Nutrition and Wellness Research Center, Ames, Iowa, United States

REFERENCES:
- [Derived] Ye Z, Arumugam V, Haugabrooks E, Williamson P, Hendrich S. Soluble dietary fiber (Fibersol-2) decreased hunger and increased satiety hormones in humans when ingested with a meal. Nutr Res. 2015 May;35(5):393-400. doi: 10.1016/j.nutres.2015.03.004. Epub 2015 Mar 18. PMID 25823991